CLINICAL TRIAL: NCT03417830
Title: An Adaptive, Open-Label Study to Evaluate the Biodistribution of 89Zirconium-labelled GSK2398852 in the Heart and Other Organs of Patients With Transthyretin Cardiomyopathy (ATTR-CM) Using Positron Emission Tomography (PET) Imaging
Brief Title: Biodistribution of 89Zirconium-labelled GSK2398852 Using PET Imaging
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in benefit/risk profile.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 204512; 2017-002665-22 (EudraCT Number)
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Results first posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-07

CONDITIONS: Amyloidosis
Keywords: miridesap; GSK2315698; 89Zirconium labelled; Positron Emission Tomography; Transthyretin cardiomyopathy; GSK2398852; dezamizumab
MeSH Terms: conditions — Amyloidosis | interventions — miridesap; dezamizumab

STUDY DESIGN:
Intervention Model Description: Part A of the study will include 3 subjects with ATTR-CM who will participate in two dosing sessions and Part B of the study will include 3 subjects with ATTR-CM who will participate in one dosing session. A single dosing session will constitute treatment with carboxy pyrrolidine hexanoyl pyrrolidine carboxylate (CPHPC), total mass dose (TMD) administration of anti-serum amyloid P (SAP) monoclonal antibody (mAb) consisting of in vivo mixing of a single infusion of unlabeled anti-SAP mAb and a separate infusion of 89Zr-GSK2398852 via a different peripheral venous line, and up to 3 serial PET scanning procedures after administration of 89Zr-GSK2398852.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects with ATTR-CM in Part A (Experimental): Approximately 3 subjects with either wild type or inherited ATTR-CM will be included. Subjects in Part A will participate in two anti-SAP dosing sessions approximately 26 days in duration. The first two subjects in Part A will have up to three 89Zr PET scans, while the remaining subject will undergo up to two 89Zr PET scans.
  Interventions: Drug: GSK2315698 (CPHPC); Drug: GSK2398852 (unlabeled anti-SAP mAb); Drug: 89Zr-GSK2398852 (89Zr-labeled anti-SAP mAb)
- Subjects with ATTR-CM in Part B (Experimental): Approximately 3 subjects with either wild type or inherited ATTR-CM will be included. Subjects in Part B will participate in one anti-SAP dosing session. Subjects will undergo up to two 89Zr PET scans.
  Interventions: Drug: GSK2315698 (CPHPC); Drug: GSK2398852 (unlabeled anti-SAP mAb); Drug: 89Zr-GSK2398852 (89Zr-labeled anti-SAP mAb)

INTERVENTIONS:
Drug: GSK2315698 (CPHPC) — GSK2315698 will be administered as 20 milligrams per hour (20 mg/hour) IV infusion (in the vein) for up to 72 hours followed by 60 milligrams (mg) three times daily as SC injection for 8 days. Dose level and frequency will be adjusted according to renal function.
  Other Names: miridesap
Drug: GSK2398852 (unlabeled anti-SAP mAb) — Subjects will be administered up to 490 mg of GSK2398852, IV. Dose level will be adjusted based on emerging imaging data.
  Other Names: dezamizumab
Drug: 89Zr-GSK2398852 (89Zr-labeled anti-SAP mAb) — 89Zr-GSK2398852 will be available as solution containing 10 mg 89Zr-GSK2398852 for Infusion. Subjects will be administered 37 (Megabecquerel) MBq radioactive dose of 89Zr-GSK2398852 by the IV route at each dosing session.

SUMMARY:
The principal aim of this study is to investigate the cardiac uptake of 89Zr-GSK2398852 in subjects with transthyretin cardiomyopathy amyloidosis (ATTR-CM), and its biodistribution to other organs. Low doses of GSK2398852 will be co-administered at levels not high enough for therapeutic benefit. This study will be conducted in two parts: Part A and Part B. Subjects in Part A will participate in up to two dosing sessions and subjects in Part B will participate in one dosing session. Subjects will undergo up to 3 PET scans at varying intervals after 89Zr-GSK2398852 administration. The total duration of study will be approximately 3 to 4 months for subjects in Part A and approximately 2 months for subjects in Part B. Part B of the study will be triggered based on data obtained in Part A and other emerging data.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 65 to 80 years of age inclusive, at the time of signing the informed consent.
* Subjects with a diagnosis of ATTR-CM: a) Wild-type ATTR status must be confirmed by genotyping and have one of the following: i) Definite histochemical identification of amyloid by Congo red staining and green birefringence in crossed polarized light in cardiac or other tissue biopsy and identification of Transthyretin amyloidosis (TTR) as the amyloid fibril protein either by immunohistochemistry or proteomic analysis OR ii) Scintigraphy Technetium-99m-labeled 3,3-diphosphono-1,2-propanodicarboxylic acid (99mTc-DPD) with confirmed myocardial uptake. b) Hereditary ATTR amyloidosis (example, TTR Val30Met) should have a known amyloidogenic TTR mutation demonstrated by genotyping and is recognized to be primarily associated with cardiomyopathy and one of the following: i) Definite histochemical identification of amyloid by Congo red staining and green birefringence in crossed polarized light in cardiac or other tissue biopsy and identification of TTR as the amyloid fibril protein either by immunohistochemistry or proteomic analysis. ii) Scintigraphy: 99mTc-DPD with confirmed myocardial uptake.
* Both male and female subjects are eligible to participate. a) Male subjects: A male subject must agree to use contraception during the treatment period and for at least 3 months after the last scan and refrain from donating sperm during this period. b) Female subjects: A female subject is eligible to participate if she is not of childbearing potential.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.
* New York Heart Association (NYHA) up to class 3; subjects should be clinically stable for at least 3 months preceding to Screening.

Exclusion Criteria:

* Cardiomyopathy primarily caused by non-amyloid diseases (example, ischemic heart disease; valvular heart disease).
* Interval from the Q wave on the ECG to point T using Fredericia's formula (QTcF) >500 milliseconds (msec).
* Sustained (at a rate of >=120 beats per minute for >=30 seconds), or symptomatic monomorphic ventricular tachycardia (VT), or rapid polymorphic VT, at Screening/Baseline cardiac monitoring.
* Systolic blood pressure <=100 millimeters of mercury (mm/Hg) based on triplicate readings at Screening.
* Unstable heart failure defined as emergency hospitalization for worsening, or decompensated heart failure, or syncopal episode within 1 month of screening.
* Implantable cardiac defibrillator (ICD) or permanent pacemaker (PPM) at Screening.
* Estimated Glomerular filtration rate (eGFR) at Screening <50 milliliters per minute (mL/min) calculated using modification of diet in renal disease (MDRD).
* Any active and persistent dermatological condition, which in the opinion of the Investigator and Medical Monitor would preclude safe participation.
* History of allogeneic stem cell transplantation, prior solid organ transplant, or anticipated to undergo solid organ transplantation, or left ventricular assist device (LVAD) implantation.
* Malignancy within last 5 years, except for basal or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix that has been successfully treated.
* Acute coronary syndrome, or any form of coronary revascularization procedure (including coronary artery bypass grafting [CABG]), within 6 months of screening.
* Symptomatic, clinically significant autonomic neuropathy which the Principal Investigator (PI) feels will preclude administration of study treatment.
* Uncontrolled hypertension during Screening.
* ALT >3 times upper limit of normal (ULN) OR bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Peripheral edema at Screening that in the opinion of the PI or designee might prevent adequate absorption of subcutaneously administered CPHPC.
* Presence of any co-morbid (example, steroid refractory rheumatoid arthritis), or an uncontrolled medical condition (example, diabetes mellitus), which in the opinion of the investigator would increase the potential risk to the subject. Investigator should liaise with the Medical Monitor where there is uncertainty as to the eligibility of a subject.
* Positive test for hepatitis B, hepatitis C and/or human immunodeficiency virus (HIV) during Screening, or within 3 months prior to first dose of study treatment.
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A [IgA] dermatosis, toxic epidermal necrolysis and exfoliative dermatitis).
* Inability to comprehend and/or understand the study patient information sheet, and/or unwillingness or inability to follow the procedures outlined in the protocol.
* Has any of the following: a) Fulfillment of diagnostic criteria for Amyloid Light-chain (AL) amyloidosis. b) Fulfillment of diagnostic criteria for amyloid A (AA) or non-TTR hereditary amyloidosis.
* ATTR Disease Load: c) Histologically proven or clinically suspected gastrointestinal TTR amyloidosis; d) Diffuse skeletal muscle uptake of 99m(Tc)-DPD on Single-photon emission computed tomography (SPECT) imaging (where available); e) Peripheral neuropathy causing more than mild morbidity (example, walking disability; neuropathic pain affecting activities of daily living); f) Proven or clinically suspected intracranial TTR involvement including ophthalmological disease.
* Non-amyloidosis related chronic liver disease (with the exception of Gilbert's syndrome or clinically asymptomatic gallstones).
* Participation in a separate clinical trial involving CPHPC within 3 months of Screening.
* Any prohibited concomitant medication within referenced timeframe.
* Treatment with another investigational drug, biological agent, or device within 6 months of screening, or 5 half-lives of the study agent, whichever is longer.
* Orthopnea of sufficient severity to preclude supine scanning as determined at Screening.
* Inability to fit inside scanner due to body size (girth).
* History of claustrophobia.
* Contraindication to magnetic resonance imaging (MRI) contrast agents.
* Contraindication for MRI scanning (as assessed by local MRI safety questionnaire), which includes but is not limited to: a) Intracranial aneurysm clips (except Sugita) or other metallic objects; b) Intra-orbital metal fragments that have not been removed; c) Pacemakers or other implanted cardiac rhythm management/monitoring devices and non-magnetic resonance (MR) conditional heart valves; d) Inner ear implants.
* Donation of blood or blood products in excess of 500 milliliters (mL) within 84 days of Screening.
* Poor or unsuitable venous access.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Wechalekar A, Antoni G, Al Azzam W, Bergstrom M, Biswas S, Chen C, Cheriyan J, Cleveland M, Cookson L, Galette P, Janiczek RL, Kwong RY, Lukas MA, Millns H, Richards D, Schneider I, Solomon SD, Sorensen J, Storey J, Thompson D, van Dongen G, Vugts DJ, Wall A, Wikstrom G, Falk RH. Pharmacodynamic evaluation and safety assessment of treatment with antibodies to serum amyloid P component in patients with cardiac amyloidosis: an open-label Phase 2 study and an adjunctive immuno-PET imaging study. BMC Cardiovasc Disord. 2022 Feb 13;22(1):49. doi: 10.1186/s12872-021-02407-6. PMID 35152886

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two part study. Part A contains two dosing sessions and Part B contain single dosing session. This study was conducted at a single center in Sweden from 06-April-18 to 20-July-2018.
Pre-assignment Details: Two participants were enrolled in Part A. The study was terminated by sponsor due to a change in the benefit:risk profile of GSK2315698+GSK2398852 (anti-serum amyloid P component [SAP] treatment) during Part A; hence, no participants were enrolled in Part B.
Groups:
- Part A: Anti-SAP: Participants with either wild type or inherited transthyretin amyloidosis restrictive cardiomyopathy (ATTR-CM) were included. Participants underwent two dosing sessions. In each dosing session, participants were administered (dependent on renal function) 20 milligram (mg) per hour or 10 mg/hour GSK2315698 for 48 hours by one intravenous infusion; followed by administration of 70 mg(session1) or 490mg (session2) GSK2398852 (unlabelled anti-SAP mAb) together with 10 mg of 89Zr-GSK2398852 (up to 37 megabecquerel of radioactive dose) via two separate intravenous infusion on Day 3. Participants also received a subcutaneous injection of GSK2315698 60 mg thrice daily for up to 8 days after administration of unlabelled anti-SAP mAb dose. Up to 3 positron emission tomography (PET) scans were performed after the end of 89Zr-GSK2398852 infusion. There was a minimum of 4 weeks of duration between dosing sessions of anti-SAP mAb.
- Part B: Anti-SAP: Participants with either wild type or ATTR-CM were planned to undergo one dosing sessions. Participants were planned to be administered 200 mg/mL GSK2315698 via intravenous infusion for 48 hours followed by administration of 100 mg/mL GSK2398852 (unlabelled anti-SAP mAb) together with 10 mg of 89Zr-GSK2398852 (up to 37 megabecquerel of radioactive dose) via two separate intravenous infusion on Day 3. Participants were planned to receive a subcutaneous injection of GSK2315698 thrice daily for up to 8 days after administration of unlabelled anti-SAP mAb dose. Up to 2 PET scans were planned to be performed after the end of 89Zr-GSK2398852 infusion.
Period: Part A (up to 26 Days)
Arm/Group | Part A: Anti-SAP | Part B: Anti-SAP
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Study Closed/Terminated | 1 | 0
Period: Part B (up to 26 Days)
Arm/Group | Part A: Anti-SAP | Part B: Anti-SAP
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated by sponsor due to a change in the benefit:risk profile of GSK2315698+GSK2398852 (anti-SAP treatment) during Part A; hence, no participants were enrolled in Part B.
Groups:
- Part A: Anti-SAP: Participants with either wild type or ATTR-CM were included. Participants underwent two dosing sessions. In each dosing session, participants were administered (dependent on renal function) 20 mg per hour or 10 mg/hour GSK2315698 for 48 hours by one intravenous infusion; followed by administration of 70 mg (session1) or 490mg (session2) GSK2398852 (unlabelled anti-SAP mAb) together with 10 mg of 89Zr-GSK2398852 (up to 37 megabecquerel of radioactive dose) via two separate intravenous infusion on Day 3. Participants also received a subcutaneous injection of GSK2315698 60 mg thrice daily for up to 8 days after administration of unlabelled anti-SAP mAb dose. Up to 3 PET scans were performed after the end of 89Zr-GSK2398852 infusion. There was a minimum of 4 weeks of duration between dosing sessions of anti-SAP mAb.
- Total: Total of all reporting groups
Arm/Group | Part A: Anti-SAP | Part B: Anti-SAP | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.5 (3.54) |  | 77.5 (3.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 1 |  | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Part A- Session 1: Peak Standardized Uptake Values (SUV) in Focal Anatomical Regions of the Heart Following 80-200 mg Dose of Anti-SAP mAb
Description: SUV was measured radioactivity concentration corrected for radioactive decay and normalized for administered amount of radioactivity per body weight. SUV was analyzed for each region of interest such as blood pool left atrium, blood pool left ventricle, blood pool right ventricle, left ventricle wall - high uptake, left ventricle wall - low uptake, mid septum - high uptake and mid septum - low uptake. Peak SUV values derived from PET images has been presented. All treated population consisted of all participants who received at least one Anti-SAP treatment including 89Zr-GSK2398852.
Time Frame: Session 1: Days 4, 5, 6 and 8
Population: All treated Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Groups:
- Part A: Anti-SAP- Session 1: Participants with either wild type or inherited ATTR-CM were included. In dosing session 1, participants were administered (dependent on renal function) 20 mg/hour or 10 mg/hour GSK2315698 for 48 hours by one intravenous infusion; followed by administration of 70 mg (session 1) GSK2398852 (unlabelled anti-SAP mAb) together with 10 mg of 89Zr-GSK2398852 (up to 37 megabecquerel of radioactive dose) via intravenous infusion on Day 3. Participants also received a subcutaneous injection of GSK2315698 60 mg thrice daily for up to 8 days after administration of unlabelled anti-SAP mAb dose. Up to 3 PET scans were performed after the end of 89Zr-GSK2398852 infusion.
Arm/Group | Part A: Anti-SAP- Session 1
Number analyzed (Participants) | 2
Grams per milliliter
  Session1:Blood pool left atrium,Day4,n=2 | 2.995 (1.4637)
  Session1:Blood pool left atrium,Day5,n=1: number analyzed (Participants) | 1
  Session1:Blood pool left atrium,Day5,n=1 | 0.550 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Blood pool left atrium,Day6,n=1: number analyzed (Participants) | 1
  Session1:Blood pool left atrium,Day6,n=1 | 0.640 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Blood pool left atrium,Day8,n=1: number analyzed (Participants) | 1
  Session1:Blood pool left atrium,Day8,n=1 | 0.400 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Blood pool left ventricle,Day4,n=2 | 2.800 (1.5274)
  Session1:Blood pool left ventricle,Day5,n=1: number analyzed (Participants) | 1
  Session1:Blood pool left ventricle,Day5,n=1 | 0.510 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Blood pool left ventricle,Day6,n=1: number analyzed (Participants) | 1
  Session1:Blood pool left ventricle,Day6,n=1 | 0.850 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Blood pool left ventricle,Day8,n=1: number analyzed (Participants) | 1
  Session1:Blood pool left ventricle,Day8,n=1 | 0.430 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Blood pool right ventricle,Day4,n=2 | 3.165 (1.1526)
  Session1:Blood pool right ventricle,Day5,n=1: number analyzed (Participants) | 1
  Session1:Blood pool right ventricle,Day5,n=1 | 1.050 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Blood pool right ventricle,Day6,n=1: number analyzed (Participants) | 1
  Session1:Blood pool right ventricle,Day6,n=1 | 0.950 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Blood pool right ventricle,Day8,n=1: number analyzed (Participants) | 1
  Session1:Blood pool right ventricle,Day8,n=1 | 1.240 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Left ventricle wall-high uptake,Day4,n=2 | 2.380 (1.4425)
  Session1:Left ventricle wall-high uptake,Day5,n=1: number analyzed (Participants) | 1
  Session1:Left ventricle wall-high uptake,Day5,n=1 | 1.290 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Left ventricle wall-high uptake,Day6,n=1: number analyzed (Participants) | 1
  Session1:Left ventricle wall-high uptake,Day6,n=1 | 3.400 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Left ventricle wall-high uptake,Day8,n=1: number analyzed (Participants) | 1
  Session1:Left ventricle wall-high uptake,Day8,n=1 | 1.440 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Left ventricle wall-low uptake,Day4,n=2 | 1.740 (1.4425)
  Session1:Left ventricle wall-low uptake,Day5,n=1: number analyzed (Participants) | 1
  Session1:Left ventricle wall-low uptake,Day5,n=1 | 0.700 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Left ventricle wall-low uptake,Day6,n=1: number analyzed (Participants) | 1
  Session1:Left ventricle wall-low uptake,Day6,n=1 | 1.840 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Left ventricle wall-low uptake,Day8,n=1: number analyzed (Participants) | 1
  Session1:Left ventricle wall-low uptake,Day8,n=1 | 0.760 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Mid septum-high uptake,Day4,n=2 | 2.335 (1.2516)
  Session1: Mid septum-high uptake,Day5,n=1: number analyzed (Participants) | 1
  Session1: Mid septum-high uptake,Day5,n=1 | 1.420 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Mid septum-high uptake,Day6,n=1: number analyzed (Participants) | 1
  Session1: Mid septum-high uptake,Day6,n=1 | 2.880 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Mid septum-high uptake,Day8,n=1: number analyzed (Participants) | 1
  Session1: Mid septum-high uptake,Day8,n=1 | 1.520 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Mid septum-low uptake,Day4,n=2 | 1.955 (1.6051)
  Session1: Mid septum-low uptake,Day5,n=1: number analyzed (Participants) | 1
  Session1: Mid septum-low uptake,Day5,n=1 | 0.780 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Mid septum-low uptake,Day6,n=1: number analyzed (Participants) | 1
  Session1: Mid septum-low uptake,Day6,n=1 | 2.230 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Mid septum-low uptake,Day8,n=1: number analyzed (Participants) | 1
  Session1: Mid septum-low uptake,Day8,n=1 | 0.610 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

2. Primary Outcome: Part A- Session 2: Peak SUV in Focal Anatomical Regions of the Heart Following Anti-SAP mAb Dose Between 200 mg and <=500 mg
Description: SUV was measured radioactivity concentration corrected for radioactive decay and normalized for administered amount of radioactivity per body weight. SUV was analyzed for each region of interest such as blood pool left atrium, blood pool left ventricle, blood pool right ventricle, left ventricle wall - high uptake, left ventricle wall - low uptake, mid septum - high uptake and mid septum - low uptake. Peak SUV values derived from PET images has been presented.
Time Frame: Session 2: Days 3, 4 and 5
Population: All treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Groups:
- Part A: Anti-SAP- Session 2: Participants with either wild type or inherited ATTR-CM were included. In dosing session 2, participants were administered (dependent on renal function) 20 mg/hour or 10 mg/hour GSK2315698 for 48 hours by one intravenous infusion; followed by administration of 490 mg (session 2) GSK2398852 (unlabelled anti-SAP mAb) together with 10 mg of 89Zr-GSK2398852 (up to 37 megabecquerel of radioactive dose) via intravenous infusion on Day 3. Participants also received a subcutaneous injection of GSK2315698 60 mg thrice daily for up to 8 days after administration of unlabelled anti-SAP mAb dose. Up to 3 PET scans were performed after the end of 89Zr-GSK2398852 infusion.
Arm/Group | Part A: Anti-SAP- Session 2
Number analyzed (Participants) | 1
Grams per milliliter
  Session2:Blood pool left atrium,Day3 | 10.290 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Blood pool left atrium,Day4 | 5.330 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Blood pool left atrium,Day5 | 3.550 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Blood pool left ventricle,Day3 | 10.120 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Blood pool left ventricle,Day4 | 4.910 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Blood pool left ventricle,Day5 | 3.110 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Blood pool right ventricle,Day3 | 10.390 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Blood pool right ventricle,Day4 | 5.160 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Blood pool right ventricle,Day5 | 3.500 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Left ventricle wall-high uptake,Day3 | 1.150 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Left ventricle wall-high uptake,Day4 | 4.540 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Left ventricle wall-high uptake,Day5 | 5.360 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Left ventricle wall-low uptake,Day3 | 3.110 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Left ventricle wall-low uptake,Day4 | 3.650 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Left ventricle wall-low uptake,Day5 | 3.980 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Mid septum-high uptake,Day3 | 4.680 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Mid septum-high uptake,Day4 | 4.200 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Mid septum-high uptake,Day5 | 4.780 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Mid septum-low uptake,Day3 | 3.580 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Mid septum-low uptake,Day4 | 3.570 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Mid septum-low uptake,Day5 | 3.800 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

3. Primary Outcome: Part B: Peak SUV in Focal Anatomical Regions of the Heart Following 80-200 mg Dose of Anti-SAP mAb
Description: SUV in focal anatomical regions of the heart was planned to be measured.
Time Frame: Days 3, 4 and 6
Population: All treated Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

4. Primary Outcome: Part B: Peak SUV in Focal Anatomical Regions of the Heart Following Anti-SAP mAb Dose Between 200 mg and <=500 mg
Description: SUV in focal anatomical regions of the heart was planned to be measured.
Time Frame: Days 3, 4 and 6
Population: All treated Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

5. Primary Outcome: Part A- Session 1: Mean SUV of Whole Heart Following 80-200 mg Dose of Anti-SAP mAb
Description: SUV was measured radioactivity concentration corrected for radioactive decay and normalized for administered amount of radioactivity per body weight.
Time Frame: Session 1: Days 4, 5, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Part A: Anti-SAP- Session 1
Number analyzed (Participants) | 2
Grams per milliliter
  Session 1: Day 4, n=2 | 2.470 (1.1738)
  Session 1: Day 5, n=1: number analyzed (Participants) | 1
  Session 1: Day 5, n=1 | 1.130 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Day 6, n=1: number analyzed (Participants) | 1
  Session 1: Day 6, n=1 | 1.320 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Day 8, n=1: number analyzed (Participants) | 1
  Session 1: Day 8, n=1 | 0.960 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

6. Primary Outcome: Part A- Session 2: Mean SUV of Whole Heart Following Anti-SAP mAb Dose Between 200 mg and <=500 mg
Description: as for outcome 5
Time Frame: Session 2: Days 3, 4 and 5
Population: All treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Part A: Anti-SAP- Session 2
Number analyzed (Participants) | 1
Grams per milliliter
  Session 2: Day 3 | 7.090 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 4 | 4.440 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 5 | 3.390 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

7. Primary Outcome: Part B: Mean SUV of Whole Heart Following 80-200 mg Dose of Anti-SAP mAb
Description: SUV of whole heart was planned to be measured.
Time Frame: Days 3, 4 and 6
Population: All treated Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

8. Primary Outcome: Part B: Mean SUV of Whole Heart Following Anti-SAP mAb Dose Between 200 mg and <=500 mg
Description: SUV of whole heart was planned to be measured.
Time Frame: Days 3, 4 and 6
Population: All treated Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

9. Secondary Outcome: Part A- Session 1: Mean SUV of Focal Radioactivity Uptake After 80-200 mg Dose of Anti-SAP mAb
Description: SUV was measured radioactivity concentration corrected for radioactive decay and normalized for administered amount of radioactivity per body weight. SUV was analyzed for each region of interest such as abdominal skin and skin of the back. Mean SUV derived from PET images has been presented.
Time Frame: Session 1: Days 4, 5, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Part A: Anti-SAP- Session 1
Number analyzed (Participants) | 2
Grams per milliliter
  Session1:Abdominal skin,Day 4,n=2 | 0.325 (0.2475)
  Session1:Abdominal skin,Day 5,n=1: number analyzed (Participants) | 1
  Session1:Abdominal skin,Day 5,n=1 | 0.080 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Abdominal skin,Day 6,n=1: number analyzed (Participants) | 1
  Session1:Abdominal skin,Day 6,n=1 | 0.940 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Abdominal skin,Day 8,n=1: number analyzed (Participants) | 1
  Session1:Abdominal skin,Day 8,n=1 | 0.140 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Skin of the back,Day 4,n=2 | 0.125 (0.1061)
  Session1:Skin of the back,Day 5,n=1: number analyzed (Participants) | 1
  Session1:Skin of the back,Day 5,n=1 | 0.060 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Skin of the back,Day 6,n=1: number analyzed (Participants) | 1
  Session1:Skin of the back,Day 6,n=1 | 0.230 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Skin of the back,Day 8,n=1: number analyzed (Participants) | 1
  Session1:Skin of the back,Day 8,n=1 | 0.100 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

10. Secondary Outcome: Part A- Session 1: Mean SUV of Focal Radioactivity Uptake After 80-200 mg Dose of Anti-SAP mAb: Thyriod Gland-goitre Hotspot
Description: SUV was measured radioactivity concentration corrected for radioactive decay and normalized for administered amount of radioactivity per body weight. SUV was analyzed for thyroid gland-goitre hotspot. Mean SUV derived from PET images has been presented.
Time Frame: Session 1: Days 4 and 6
Population: All treated Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Part A: Anti-SAP- Session 1
Number analyzed (Participants) | 2
Grams per milliliter
  Session 1: Day 4: number analyzed (Participants) | 1
  Session 1: Day 4 | 4.670 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Day 6: number analyzed (Participants) | 1
  Session 1: Day 6 | 4.240 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

11. Secondary Outcome: Part A- Session 2: Mean SUV of Focal Radioactivity Uptake After Anti-SAP mAb Dose Between 200 mg and <=500 mg
Description: SUV was measured radioactivity concentration corrected for radioactive decay and normalized for administered amount of radioactivity per body weight. SUV was analyzed for each region of interest such as thyroid gland-goitre hotspot, abdominal skin and skin of the back. Mean SUV derived from PET images has been presented.
Time Frame: Session 2: Days 3, 4 and 5
Population: All treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Part A: Anti-SAP- Session 2
Number analyzed (Participants) | 1
Grams per milliliter
  Session2:Thyroid gland-goitre hotspot,Day 3 | 1.890 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Thyroid gland-goitre hotspot,Day 4 | 3.690 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Thyroid gland-goitre hotspot,Day 5 | 3.190 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Abdominal skin,Day 3 | 0.620 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Abdominal skin,Day 4 | 0.780 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Abdominal skin,Day 5 | 0.870 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Skin of the back,Day 3 | 0.220 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Skin of the back,Day 4 | 0.250 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Skin of the back,Day 5 | 0.330 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

12. Secondary Outcome: Part B: Mean SUV of Focal Radioactivity Uptake After 80-200 mg Dose of Anti-SAP mAb
Description: SUV of focal radioactivity uptake for different organs/tissues was planned to be measured.
Time Frame: Days 3, 4 and 6
Population: All treated Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

13. Secondary Outcome: Part B: Mean SUV of Focal Radioactivity Uptake After Anti-SAP mAb Dose Between 200 mg and <=500 mg
Description: SUV of focal radioactivity uptake for different organs/tissues was planned to be measured.
Time Frame: Days 3, 4 and 6
Population: All treated Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

14. Secondary Outcome: Part A- Session 1: Mean SUV of Total Radioactivity Uptake After 80-200 mg Dose of Anti-SAP mAb
Description: SUV was measured radioactivity concentration corrected for radioactive decay and normalized for administered amount of radioactivity per body weight. SUV was analyzed for each region of interest such as adrenal gland, aorta, bone marrow, kidney, liver, spleen, abdominal region, brain, lung, parotid gland, and thigh. Mean SUV derived from PET images has been presented.
Time Frame: Session 1: Days 4, 5, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Part A: Anti-SAP- Session 1
Number analyzed (Participants) | 2
Grams per milliliter
  Session1:Adrenal gland,Day 4,n=2 | 11.665 (1.9304)
  Session1:Adrenal gland,Day 5,n=1: number analyzed (Participants) | 1
  Session1:Adrenal gland,Day 5,n=1 | 10.770 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Adrenal gland,Day 6,n=1: number analyzed (Participants) | 1
  Session1:Adrenal gland,Day 6,n=1 | 12.020 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Adrenal gland,Day 8,n=1: number analyzed (Participants) | 1
  Session1:Adrenal gland,Day 8,n=1 | 10.900 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Aorta,Day 4,n=2 | 2.580 (1.3859)
  Session1: Aorta,Day 5,n=1: number analyzed (Participants) | 1
  Session1: Aorta,Day 5,n=1 | 0.360 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Aorta,Day 6,n=1: number analyzed (Participants) | 1
  Session1: Aorta,Day 6,n=1 | 0.500 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Aorta,Day 8,n=1: number analyzed (Participants) | 1
  Session1: Aorta,Day 8,n=1 | 0.650 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Bone marrow,Day 4,n=2 | 3.015 (0.7990)
  Session1: Bone marrow,Day 5,n=1: number analyzed (Participants) | 1
  Session1: Bone marrow,Day 5,n=1 | 3.170 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Bone marrow,Day 6,n=1: number analyzed (Participants) | 1
  Session1: Bone marrow,Day 6,n=1 | 2.210 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Bone marrow,Day 8,n=1: number analyzed (Participants) | 1
  Session1: Bone marrow,Day 8,n=1 | 3.880 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Kidney,Day 4,n=2 | 4.910 (1.1738)
  Session1: Kidney,Day 5,n=1: number analyzed (Participants) | 1
  Session1: Kidney,Day 5,n=1 | 5.130 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Kidney,Day 6,n=1: number analyzed (Participants) | 1
  Session1: Kidney,Day 6,n=1 | 3.840 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Kidney,Day 8,n=1: number analyzed (Participants) | 1
  Session1: Kidney,Day 8,n=1 | 4.820 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Liver,Day 4,n=2 | 17.805 (6.8519)
  Session1:Liver,Day 5,n=1: number analyzed (Participants) | 1
  Session1:Liver,Day 5,n=1 | 25.560 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Liver,Day 6,n=1: number analyzed (Participants) | 1
  Session1:Liver,Day 6,n=1 | 16.940 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Liver,Day 8,n=1: number analyzed (Participants) | 1
  Session1:Liver,Day 8,n=1 | 24.800 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Spleen,Day 4,n=2 | 11.425 (2.2981)
  Session1: Spleen,Day 5,n=1: number analyzed (Participants) | 1
  Session1: Spleen,Day 5,n=1 | 11.050 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Spleen,Day 6,n=1: number analyzed (Participants) | 1
  Session1: Spleen,Day 6,n=1 | 10.060 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Spleen,Day 8,n=1: number analyzed (Participants) | 1
  Session1: Spleen,Day 8,n=1 | 11.340 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Abdominal region,Day 4,n=2 | 1.070 (0.5374)
  Session1:Abdominal region,Day 5,n=1: number analyzed (Participants) | 1
  Session1:Abdominal region,Day 5,n=1 | 0.610 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Abdominal region,Day 6,n=1: number analyzed (Participants) | 1
  Session1:Abdominal region,Day 6,n=1 | 1.740 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Abdominal region,Day 8,n=1: number analyzed (Participants) | 1
  Session1:Abdominal region,Day 8,n=1 | 0.460 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Brain,Day 4,n=2 | 0.125 (0.0354)
  Session1: Brain,Day 5,n=1: number analyzed (Participants) | 1
  Session1: Brain,Day 5,n=1 | 0.060 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Brain,Day 6,n=1: number analyzed (Participants) | 1
  Session1: Brain,Day 6,n=1 | 0.070 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Brain,Day 8,n=1: number analyzed (Participants) | 1
  Session1: Brain,Day 8,n=1 | 0.070 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Lung,Day 4,n=2 | 0.555 (0.1202)
  Session1: Lung,Day 5,n=1: number analyzed (Participants) | 1
  Session1: Lung,Day 5,n=1 | 0.440 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Lung,Day 6,n=1: number analyzed (Participants) | 1
  Session1: Lung,Day 6,n=1 | 0.260 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Lung,Day 8,n=1: number analyzed (Participants) | 1
  Session1: Lung,Day 8,n=1 | 0.400 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Parotid gland,Day 4,n=2 | 0.570 (0.2970)
  Session1:Parotid gland,Day 5,n=1: number analyzed (Participants) | 1
  Session1:Parotid gland,Day 5,n=1 | 0.240 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Parotid gland,Day 6,n=1: number analyzed (Participants) | 1
  Session1:Parotid gland,Day 6,n=1 | 0.580 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1:Parotid gland,Day 8,n=1: number analyzed (Participants) | 1
  Session1:Parotid gland,Day 8,n=1 | 0.170 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Thigh,Day 4,n=2 | 0.260 (0.1131)
  Session1: Thigh,Day 5,n=1: number analyzed (Participants) | 1
  Session1: Thigh,Day 5,n=1 | 0.110 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Thigh,Day 6,n=1: number analyzed (Participants) | 1
  Session1: Thigh,Day 6,n=1 | 0.200 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Thigh,Day 8,n=1: number analyzed (Participants) | 1
  Session1: Thigh,Day 8,n=1 | 0.110 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

15. Secondary Outcome: Part A- Session 1: Mean SUV of Total Radioactivity Uptake After 80-200 mg Dose of Anti-SAP mAb: Thyroid Gland-goitre
Description: SUV was measured radioactivity concentration corrected for radioactive decay and normalized for administered amount of radioactivity per body weight. SUV was analyzed for thyroid gland-goitre. Mean SUV derived from PET images has been presented.
Time Frame: Session 1: Days 4 and 6
Population: All treated Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Part A: Anti-SAP- Session 1
Number analyzed (Participants) | 2
Grams per milliliter
  Session1: Day 4: number analyzed (Participants) | 1
  Session1: Day 4 | 1.630 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Day 6: number analyzed (Participants) | 1
  Session1: Day 6 | 1.390 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

16. Secondary Outcome: Part A- Session 1: Mean SUV of Total Radioactivity Uptake After 80-200 mg Dose of Anti-SAP mAb: Testes
Description: SUV was measured radioactivity concentration corrected for radioactive decay and normalized for administered amount of radioactivity per body weight. SUV was analyzed for testes. Mean SUV derived from PET images has been presented.
Time Frame: Session 1: Days 4, 5 and 8
Population: All treated Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Part A: Anti-SAP- Session 1
Number analyzed (Participants) | 1
Grams per milliliter
  Session1: Day 4 | 5.400 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Day 5 | 5.520 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session1: Day 8 | 5.670 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

17. Secondary Outcome: Part A- Session 2: Mean SUV of Total Radioactivity Uptake After Anti-SAP mAb Dose Between 200 mg and <=500 mg
Description: SUV was measured radioactivity concentration corrected for radioactive decay and normalized for administered amount of radioactivity per body weight. SUV was analyzed for each region of interest such as adrenal gland, aorta, bone marrow, kidney, liver, spleen, abdominal region, brain, lung, parotid gland, thigh, and thyroid gland- goitre. Mean SUV derived from PET images has been presented.
Time Frame: Session 2: Days 3, 4, and 5
Population: All treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Part A: Anti-SAP- Session 2
Number analyzed (Participants) | 1
Grams per milliliter
  Session2: Adrenal gland,Day 3 | 4.800 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Adrenal gland,Day 4 | 8.380 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Adrenal gland,Day 5 | 6.360 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Aorta,Day 3 | 10.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Aorta,Day 4 | 5.890 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Aorta,Day 5 | 3.310 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Bone marrow,Day 3 | 1.860 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Bone marrow,Day 4 | 1.910 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Bone marrow,Day 5 | 1.410 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Kidney,Day 3 | 2.700 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Kidney,Day 4 | 3.260 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Kidney,Day 5 | 2.890 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Liver,Day 3 | 4.770 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Liver,Day 4 | 7.560 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Liver,Day 5 | 8.340 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Spleen,Day 3 | 4.440 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Spleen,Day 4 | 5.140 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Spleen,Day 5 | 5.440 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Abdominal region,Day 3 | 0.900 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Abdominal region,Day 4 | 2.170 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Abdominal region,Day 5 | 2.370 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Brain,Day 3 | 0.370 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Brain,Day 4 | 0.210 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Brain,Day 5 | 0.110 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Lung,Day 3 | 1.230 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Lung,Day 4 | 0.930 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Lung,Day 5 | 0.790 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Parotid gland,Day 3 | 1.550 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Parotid gland,Day 4 | 1.180 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Parotid gland,Day 5 | 0.850 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Thigh,Day 3 | 0.630 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Thigh,Day 4 | 0.530 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2: Thigh,Day 5 | 0.330 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Thyroid gland-goitre,Day 3 | 1.870 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Thyroid gland-goitre,Day 4 | 2.090 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session2:Thyroid gland-goitre,Day 5 | 1.950 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

18. Secondary Outcome: Part B: Mean SUV of Total Radioactivity Uptake After 80-200 mg Dose of Anti-SAP mAb
Description: SUV of total radioactivity uptake for different organs/tissues was planned to be measured.
Time Frame: Days 3, 4 and 6
Population: All treated Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

19. Secondary Outcome: Part B: Mean SUV of Total Radioactivity Uptake After an Anti-SAP mAb Dose Between 200 mg and <=500 mg
Description: SUV of total radioactivity uptake for different organs/tissues was planned to be measured.
Time Frame: Days 3, 4 and 6
Population: All treated Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

20. Secondary Outcome: Part A: Maximum Concentration in Plasma (Cmax) of Total mAb
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of total mAb (unlabelled GSK2398852 and 89Zr-GSK2398852). PK Population consisted of all participants from the All Treated Population for whom a PK sample was obtained and analyzed.
Time Frame: Sessions 1 and 2: Day 3 (pre-dose, halfway infusion, end of infusion, 4 and 7 hours after end of infusion), Days 4, 5, 6 and 7
Population: PK Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Full Range); unit: Nanograms per milliliter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Nanograms per milliliter
  Session 1, n=2 | 18061.0 [7474 to 28648]
  Session 2, n=1: number analyzed (Participants) | 1
  Session 2, n=1 | 226994.0 [226994 to 226994]

21. Secondary Outcome: Part B: Cmax of Total mAb
Description: Blood samples were planned to be collected at indicated time points for PK analysis of total mAb.
Time Frame: Day 3 (pre-dose, end of infusion, 4 and 7 hours post-infusion), Days 4, 5, 6, 7 and 8
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

22. Secondary Outcome: Part A: Time Associated With Cmax (Tmax) of Total mAb
Description: Blood samples were collected at indicated time points for PK analysis of total mAb (unlabelled GSK2398852 and 89Zr-GSK2398852).
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Full Range); unit: Hours
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Hours
  Session 1, n=2 | 3.010 [1.02 to 5.00]
  Session 2, n=1: number analyzed (Participants) | 1
  Session 2, n=1 | 6.100 [6.10 to 6.10]

23. Secondary Outcome: Part B: Tmax of Total mAb
Description: Blood samples were planned to be collected at indicated time points for PK analysis of total mAb.
Time Frame: Day 3 (pre-dose, end of infusion, 4 and 7 hours post-infusion), Days 4, 5, 6, 7 and 8
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

24. Secondary Outcome: Part A: Clearance of Total mAb
Description: as for outcome 22
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Full Range); unit: Liters per hour
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Liters per hour
  Session 1, n=2 | NA [NA to NA] — Data could not be analyzed because an estimate of Clearance for Total mAb could not be derived given the observed PK profile and data below the limit of quantitation.
  Session 2, n=1: number analyzed (Participants) | 1
  Session 2, n=1 | NA [NA to NA] — Data could not be analyzed because an estimate of Clearance for Total mAb could not be derived given the observed PK profile and data below the limit of quantitation.

25. Secondary Outcome: Part B: Clearance of Total mAb
Description: Blood samples were planned to be collected at indicated time points for PK analysis of total mAb.
Time Frame: Day 3 (pre-dose, end of infusion, 4 and 7 hours post-infusion), Days 4, 5, 6, 7 and 8
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

26. Secondary Outcome: Part A: Terminal Half-life (T1/2) of Total mAb
Description: as for outcome 22
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Full Range); unit: Hours
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Hours
  Session 1, n=2 | 17.70 [13.5 to 21.9]
  Session 2, n=1: number analyzed (Participants) | 1
  Session 2, n=1 | 23.10 [23.1 to 23.1]

27. Secondary Outcome: Part B: T1/2 of Total mAb
Description: Blood samples were planned to be collected at indicated time points for PK analysis of total mAb.
Time Frame: Day 3 (pre-dose, end of infusion, 4 and 7 hours post-infusion), Days 4, 5, 6, 7 and 8
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

28. Secondary Outcome: Part A:Area Under the Concentration Time Curve Till Last Observation (AUC[0 to t]) of Total mAb
Description: as for outcome 22
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Hours*nanogram per milliliter
  Session 1, n=2 | 471241.0 [173964 to 768518]
  Session 2, n=1: number analyzed (Participants) | 1
  Session 2, n=1 | 8274231.0 [8274231 to 8274231]

29. Secondary Outcome: Part B: AUC(0 to t) of Total mAb
Description: Blood samples were planned to be collected at indicated time points for PK analysis of total mAb.
Time Frame: Day 3 (pre-dose, end of infusion, 4 and 7 hours post-infusion), Days 4, 5, 6, 7 and 8
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

30. Secondary Outcome: Part A: Area Under the Concentration Time Curve Till Time Infinity (AUC[0 to Infinity]) of Total mAb
Description: as for outcome 22
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Hours*nanogram per milliliter
  Session 1, n=2 | 487420.5 [186190 to 788651]
  Session 2, n=1: number analyzed (Participants) | 1
  Session 2, n=1 | 8696309.0 [8696309 to 8696309]

31. Secondary Outcome: Part B: AUC(0 to Infinity) of Total mAb
Description: Blood samples were planned to be collected at indicated time points for PK analysis of total mAb.
Time Frame: Day 3 (pre-dose, end of infusion, 4 and 7 hours post-infusion), Days 4, 5, 6, 7 and 8
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

32. Secondary Outcome: Part A: Cmax of 89Zr-GSK2398852 PKs of Radioactivity (Radio-PK)
Description: Blood samples were collected at indicated time points for measurement of radioactivity. Radioactivity reflected the total concentration of 89Zr-GSK2398852 and its radioactive metabolites. Plasma radioactive concentration was measured using scintillation counter.
Time Frame: Sessions 1 and 2: Day 3 (10 minutes, 60 minutes, 4 hours, 7 hours post-dose), Days 4, 5 and 6
Population: as for outcome 20
Measure: Mean (Full Range); unit: Becquerel per gram
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Becquerel per gram
  Session 1, n=2 | 9240.5 [6599 to 11882]
  Session 2, n=1: number analyzed (Participants) | 1
  Session 2, n=1 | 11923.0 [11923 to 11923]

33. Secondary Outcome: Part B: Cmax of 89Zr-GSK2398852 Radio-PK
Description: Blood samples were planned to be collected at indicated time points for measurement of radioactivity. Radioactivity reflected the total concentration of 89Zr-GSK2398852 and its radioactive metabolites. Plasma radioactive concentration was planned to be measured by scintillation counter.
Time Frame: Day 3 (10 minutes, 60 minutes, 4 hours, 7 hours post-dose), Days 4, 5 and 6
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

34. Secondary Outcome: Part A: Tmax of 89Zr- GSK2398852 Radio-PK
Description: as for outcome 32
Time Frame: Sessions 1 and 2: Day 3 (10 minutes, 60 minutes, 4 hours, 7 hours post-dose), Days 4, 5 and 6
Population: as for outcome 20
Measure: Mean (Full Range); unit: Hours
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Hours
  Session 1, n=2 | 1.160 [1.15 to 1.17]
  Session 2, n=1: number analyzed (Participants) | 1
  Session 2, n=1 | 1.100 [1.10 to 1.10]

35. Secondary Outcome: Part B: Tmax of 89Zr-GSK2398852 Radio-PK
Description: as for outcome 33
Time Frame: Day 3 (10 minutes, 60 minutes, 4 hours, 7 hours post-dose), Days 4, 5 and 6
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

36. Secondary Outcome: Part A: T1/2 of 89Zr- GSK2398852 Radio-PK
Description: as for outcome 32
Time Frame: Sessions 1 and 2: Day 3 (10 minutes, 60 minutes, 4 hours, 7 hours post-dose), Days 4, 5 and 6
Population: as for outcome 20
Measure: Mean (Full Range); unit: Hours
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Hours
  Session 1, n=2 | 14.50 [13.8 to 15.2]
  Session 2, n=1: number analyzed (Participants) | 1
  Session 2, n=1 | 26.70 [26.7 to 26.7]

37. Secondary Outcome: Part B: T1/2 of 89Zr- GSK2398852 Radio-PK
Description: as for outcome 33
Time Frame: Day 3 (10 minutes, 60 minutes, 4 hours, 7 hours post-dose), Days 4, 5 and 6
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

38. Secondary Outcome: Part A: AUC(0 to t) of 89Zr- GSK2398852 Radio-PK
Description: as for outcome 32
Time Frame: Sessions 1 and 2: Day 3 (10 minutes, 60 minutes, 4 hours, 7 hours post-dose), Days 4, 5 and 6
Population: as for outcome 20
Measure: Mean (Full Range); unit: Hours*Becquerel per gram
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Hours*Becquerel per gram
  Session 1, n=2 | 168044.5 [92052 to 244037]
  Session 2, n=1: number analyzed (Participants) | 1
  Session 2, n=1 | 386077.0 [386077 to 386077]

39. Secondary Outcome: Part B: AUC(0 to t) of 89Zr- GSK2398852 Radio-PK
Description: as for outcome 33
Time Frame: Day 3 (10 minutes, 60 minutes, 4 hours, 7 hours post-dose), Days 4, 5 and 6
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

40. Secondary Outcome: Part A: AUC(0 to Infinity) of 89Zr- GSK2398852 Radio-PK
Description: as for outcome 32
Time Frame: Sessions 1 and 2: Day 3 (10 minutes, 60 minutes, 4 hours, 7 hours post-dose), Days 4, 5 and 6
Population: as for outcome 20
Measure: Mean (Full Range); unit: Hours*Becquerel per gram
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Hours*Becquerel per gram
  Session 1, n=2 | 174764.0 [96432 to 253096]
  Session 2, n=1: number analyzed (Participants) | 1
  Session 2, n=1 | 457666.0 [457666 to 457666]

41. Secondary Outcome: Part B: AUC(0 to Infinity) of 89Zr- GSK2398852 Radio-PK
Description: as for outcome 33
Time Frame: Day 3 (10 minutes, 60 minutes, 4 hours, 7 hours post-dose), Days 4, 5 and 6
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

42. Secondary Outcome: Part A: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other important medical events which may require medical or surgical intervention. Safety Population consisted of all participants who received at least one dose of GSK2315698, GSK2398852 or 89Zr-GSK2398852.
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants
  AEs | 2
  SAEs | 0

43. Secondary Outcome: Part B: Number of Participants With AEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other important medical events which may require medical or surgical intervention.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

44. Secondary Outcome: Part A: Number of Participants With Skin Rashes
Description: Rash was graded as Grade 1 to Grade 4 based on symptoms and body surface area (BSA) affected; Grade 1: <10 percent (%) BSA and asymptomatic; Grade 2: 10-30% BSA and/or mild symptoms (pain, itch and burning); Grade 3: >30% BSA and/or moderate/severe symptoms (pain, itch and burning); and Grade 4: any rash with mucosal or systemic involvement (such as evidence of renal involvement).
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants
  Grade 1 | 0
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 0

45. Secondary Outcome: Part B: Number of Participants With Skin Rashes
Description: Rash was planned to be graded as Grade 1 to Grade 4 based on symptoms and BSA affected; Grade 1: <10% BSA and asymptomatic; Grade 2: 10-30% BSA and/or mild symptoms (pain, itch and burning); Grade 3: >30% BSA and/or moderate/severe symptoms (pain, itch and burning); and Grade 4: any rash with mucosal or systemic involvement (such as evidence of renal involvement).
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

46. Secondary Outcome: Part A: Number of Participants With Cardiac Adverse Events
Description: The number of participants with any cardiovascular AEs i.e. any AE coded to the cardiovascular system organ class are presented.
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants | 0

47. Secondary Outcome: Part B: Number of Participants With Cardiac Adverse Events
Description: The number of participants with any cardiovascular AEs i.e. any AE coded to the cardiovascular system organ class were planned to be reported.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

48. Secondary Outcome: Part A: Number of Participants With Infusion Related Reactions
Description: Number of participants with any infusion related reactions are presented.
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants | 0

49. Secondary Outcome: Part B: Number of Participants With Infusion Related Reactions
Description: Number of participants with any infusion related reactions were planned to be reported.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

50. Secondary Outcome: Part A: Change From Baseline in Cardiac Troponin T and N-terminal Prohormone of Brain Natriuretic Peptide (NT-ProBNP)
Description: Blood samples were collected to analyze the troponin T and NT-ProBNP at indicated time points. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Session 1: Baseline (Day 1 Pre-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10 and 26; Session 2: Day 1- Pre-dose, Days 2, 3, 4, 5, 6, 7, 8, 9, 10 and 26
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanograms per liter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Nanograms per liter
  Troponin T:Session1-Day2,n=2 | -6.45 (5.020)
  Troponin T:Session1-Day3,n=2 | -13.15 (13.930)
  Troponin T:Session1-Day4,n=2 | 2.40 (5.091)
  Troponin T:Session1-Day5,n=2 | -4.80 (3.111)
  Troponin T:Session1-Day6,n=2 | 0.80 (4.525)
  Troponin T:Session1-Day7,n=2 | -4.85 (3.041)
  Troponin T:Session1-Day8,n=2 | -1.45 (0.636)
  Troponin T:Session1-Day9,n=2 | -4.65 (3.323)
  Troponin T:Session1-Day10,n=2 | 17.00 (26.870)
  Troponin T:Session1-Day26,n=2 | -5.45 (5.020)
  Troponin T:Session2-Day1-pre-dose,n=1: number analyzed (Participants) | 1
  Troponin T:Session2-Day1-pre-dose,n=1 | -2.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Troponin T:Session2-Day2,n=1: number analyzed (Participants) | 1
  Troponin T:Session2-Day2,n=1 | -4.40 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Troponin T:Session2-Day3,n=1: number analyzed (Participants) | 1
  Troponin T:Session2-Day3,n=1 | -2.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Troponin T:Session2-Day4,n=1: number analyzed (Participants) | 1
  Troponin T:Session2-Day4,n=1 | -2.90 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Troponin T:Session2-Day5,n=1: number analyzed (Participants) | 1
  Troponin T:Session2-Day5,n=1 | -3.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Troponin T:Session2-Day6,n=1: number analyzed (Participants) | 1
  Troponin T:Session2-Day6,n=1 | -3.70 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Troponin T:Session2-Day7,n=1: number analyzed (Participants) | 1
  Troponin T:Session2-Day7,n=1 | -2.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Troponin T:Session2-Day8,n=1: number analyzed (Participants) | 1
  Troponin T:Session2-Day8,n=1 | -3.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Troponin T:Session2-Day9,n=1: number analyzed (Participants) | 1
  Troponin T:Session2-Day9,n=1 | -2.60 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Troponin T:Session2-Day10,n=1: number analyzed (Participants) | 1
  Troponin T:Session2-Day10,n=1 | -2.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Troponin T:Session2-Day26,n=1: number analyzed (Participants) | 1
  Troponin T:Session2-Day26,n=1 | -3.60 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  NT-ProBNP:Session1-Day2,n=2 | -525.0 (530.33)
  NT-ProBNP:Session1-Day3,n=2 | -525.0 (502.05)
  NT-ProBNP:Session1-Day4,n=2 | 835.0 (601.04)
  NT-ProBNP:Session1-Day5,n=2 | -35.0 (7.07)
  NT-ProBNP:Session1-Day6,n=2 | 360.0 (1004.09)
  NT-ProBNP:Session1-Day7,n=2 | 470.0 (636.40)
  NT-ProBNP:Session1-Day8,n=2 | 540.0 (579.83)
  NT-ProBNP:Session1-Day9,n=2 | -90.0 (381.84)
  NT-ProBNP:Session1-Day10,n=2 | 585.0 (1124.30)
  NT-ProBNP:Session1-Day26,n=2 | 115.0 (558.61)
  NT-ProBNP:Session2-Day1-pre-dose,n=1: number analyzed (Participants) | 1
  NT-ProBNP:Session2-Day1-pre-dose,n=1 | 20.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  NT-ProBNP:Session2-Day2,n=1: number analyzed (Participants) | 1
  NT-ProBNP:Session2-Day2,n=1 | -80.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  NT-ProBNP:Session2-Day3,n=1: number analyzed (Participants) | 1
  NT-ProBNP:Session2-Day3,n=1 | -240.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  NT-ProBNP:Session2-Day4,n=1: number analyzed (Participants) | 1
  NT-ProBNP:Session2-Day4,n=1 | 280.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  NT-ProBNP:Session2-Day5,n=1: number analyzed (Participants) | 1
  NT-ProBNP:Session2-Day5,n=1 | 60.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  NT-ProBNP:Session2-Day6,n=1: number analyzed (Participants) | 1
  NT-ProBNP:Session2-Day6,n=1 | 1040.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  NT-ProBNP:Session2-Day7,n=1: number analyzed (Participants) | 1
  NT-ProBNP:Session2-Day7,n=1 | 1030.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  NT-ProBNP:Session2-Day8,n=1: number analyzed (Participants) | 1
  NT-ProBNP:Session2-Day8,n=1 | 400.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  NT-ProBNP:Session2-Day9,n=1: number analyzed (Participants) | 1
  NT-ProBNP:Session2-Day9,n=1 | 120.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  NT-ProBNP:Session2-Day10,n=1: number analyzed (Participants) | 1
  NT-ProBNP:Session2-Day10,n=1 | -40.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  NT-ProBNP:Session2-Day26,n=1: number analyzed (Participants) | 1
  NT-ProBNP:Session2-Day26,n=1 | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

51. Secondary Outcome: Part B: Change From Baseline in Cardiac Troponin T and NT-ProBNP
Description: Blood samples were planned to be collected to analyze the troponin T and NT-ProBNP at indicated time points. Baseline was considered as the latest pre-dose assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline and up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

52. Secondary Outcome: Part A: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings
Description: 12-lead ECGs were measured in a semi-supine position using an automated ECG machine after approximately 5 minutes of rest for the participant. Abnormal findings were categorized as clinically significant (CS) and not clinically significant (NCS). Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants
  CS | 0
  NCS | 2

53. Secondary Outcome: Part B: Number of Participants With Abnormal 12-lead ECG Findings
Description: 12-lead ECGs were planned to be measured in a semi-supine position using an automated ECG machine after approximately 5 minutes of rest for the participant.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

54. Secondary Outcome: Part A: Number of Participants With Abnormal Inpatient Cardiac Telemetry
Description: Continuous inpatient cardiac monitoring was performed via remote cardiac telemetry device. Abnormal findings were categorized as CS and NCS. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants
  CS | 0
  NCS | 2

55. Secondary Outcome: Part B: Number of Participants With Abnormal Inpatient Cardiac Telemetry
Description: Continuous inpatient cardiac monitoring was planned to be performed via remote cardiac telemetry device.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

56. Secondary Outcome: Part A: Number of Participants With Abnormal Outpatient Cardiac Telemetry
Description: Continuous outpatient cardiac monitoring was performed via remote cardiac bodyguardian telemetry device. Abnormal findings were categorized as CS and NCS. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants
  CS | 0
  NCS | 2

57. Secondary Outcome: Part B: Number of Participants With Abnormal Outpatient Cardiac Telemetry
Description: Continuous outpatient cardiac monitoring was planned to be performed via remote cardiac bodyguardian telemetry device.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

58. Secondary Outcome: Part A: Number of Participants With Abnormal Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in a semi-supine position after 5 minutes of rest for the participant. Potential Clinical Importance (PCI) ranges for the SBP and DBP were as follows: SBP- <90 and >180 millimeters of mercury (mmHg), and DBP- <30 and >110 mmHg.
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants
  SBP | 0
  DBP | 0

59. Secondary Outcome: Part B: Number of Participants With Abnormal SBP and DBP
Description: SBP and DBP were planned to be measured in a semi-supine position after 5 minutes of rest for the participant.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

60. Secondary Outcome: Part A: Number of Participants With Abnormal Temperature
Description: Temperature was measured in a semi-supine position after 5 minutes of rest for the participant. Normal range for temperature was as follows: temperature- >37.5 degree celsius.
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants | 0

61. Secondary Outcome: Part B: Number of Participants With Abnormal Temperature
Description: Temperature was planned to be measured in a semi-supine position after 5 minutes of rest for the participant.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

62. Secondary Outcome: Part A: Number of Participants With Abnormal Respiratory Rate
Description: Respiratory rate was measured in a semi-supine position after 5 minutes of rest for the participant. Normal range for the respiratory rate was as follows: respiratory rate- <12 and >25 breaths per minute.
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants | 0

63. Secondary Outcome: Part B: Number of Participants With Abnormal Respiratory Rate
Description: Respiratory rate was planned to be measured in a semi-supine position after 5 minutes of rest for the participant.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

64. Secondary Outcome: Part A: Number of Participants With Abnormal Pulse Rate
Description: Pulse rate were measured in a semi-supine position after 5 minutes of rest for the participant. PCI range for the pulse rate was as follows: pulse rate- <35 and >140 beats per minute (bpm).
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants | 0

65. Secondary Outcome: Part B: Number of Participants With Abnormal Pulse Rate
Description: Pulse rate was planned to be measured in a semi-supine position after 5 minutes of rest for the participant.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

66. Secondary Outcome: Part A: Number of Participants With New Abnormal Physical Examination Findings
Description: A full and brief physical examination was performed, including assessments of the skin, lungs, cardiovascular system and abdomen (liver and spleen).
Time Frame: Session 1: At screening (within 35 days of Anti-SAP treatment of session 1), Day 1 Pre-dose, Day 3, Day 5, Day 8 and Day 11; Session 2: Day 1 Pre-dose, Day 3, Day 5, Day 8 and Day 11
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants
  Session 1:Screening,n=2 | 1
  Session1:Day 1 Pre-dose,n=2 | 2
  Session1:Day 3,n=2 | 0
  Session 1:Day 5,n=2 | 1
  Session1:Day 8,n=2 | 0
  Session1:Day 11,n=2 | 0
  Session2:Day 1 Pre-dose,n=1: number analyzed (Participants) | 1
  Session2:Day 1 Pre-dose,n=1 | 0
  Session2:Day 3,n=1: number analyzed (Participants) | 1
  Session2:Day 3,n=1 | 0
  Session2:Day 5,n=1: number analyzed (Participants) | 1
  Session2:Day 5,n=1 | 1
  Session2:Day 8,n=1: number analyzed (Participants) | 1
  Session2:Day 8,n=1 | 0
  Session2:Day 11,n=1: number analyzed (Participants) | 1
  Session2:Day 11,n=1 | 0

67. Secondary Outcome: Part B: Number of Participants With New Abnormal Physical Examination Findings
Description: A full and brief physical examination was planned to be performed, including assessments of the skin, lungs, cardiovascular system and abdomen (liver and spleen).
Time Frame: At screening (within 35 days of Anti-SAP treatment), Days 1, 3, 5, 8 and 11
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

68. Secondary Outcome: Part A: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: Blood samples were collected to analyze the hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelets. Baseline was considered as the latest pre-dose assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Session 1: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26; Session 2: Day 1-Pre-dose, Days 3, 5, 7, 10 and 26
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Billion cells per liter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Billion cells per liter
  Session 1: Basophils, Day 3, n=2 | 0.000 (0.0141)
  Session 1: Basophils, Day 5, n=2 | -0.010 (0.0000)
  Session 1: Basophils, Day 7, n=2 | -0.015 (0.0071)
  Session 1: Basophils, Day 10, n=2 | -0.015 (0.0071)
  Session 1: Basophils, Day 26, n=2 | -0.005 (0.0071)
  Session 2: Basophils, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Basophils, Day1-pre-dose, n=1 | -0.010 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Basophils, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Basophils, Day 3, n=1 | -0.010 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Basophils, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Basophils, Day 5, n=1 | -0.020 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Basophils, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Basophils, Day 7, n=1 | -0.010 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Basophils, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Basophils, Day 10, n=1 | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Basophils, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Basophils, Day 26, n=1 | -0.010 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Eosinophils, Day 3, n=2 | -0.025 (0.3182)
  Session 1: Eosinophils, Day 5, n=2 | 0.050 (0.2121)
  Session 1: Eosinophils, Day 7, n=2 | 0.000 (0.1414)
  Session 1: Eosinophils, Day 10, n=2 | 0.000 (0.1414)
  Session 1: Eosinophils, Day 26, n=2 | 0.050 (0.3536)
  Session 2: Eosinophils, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Eosinophils, Day1-pre-dose, n=1 | -0.100 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Eosinophils, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Eosinophils, Day 3, n=1 | -0.100 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Eosinophils, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Eosinophils, Day 5, n=1 | -0.200 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Eosinophils, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Eosinophils, Day 7, n=1 | -0.100 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Eosinophils, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Eosinophils, Day 10, n=1 | -0.100 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Eosinophils, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Eosinophils, Day 26, n=1 | -0.230 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Lymphocytes, Day 3, n=2 | -0.05 (0.636)
  Session 1: Lymphocytes, Day 5, n=2 | 0.30 (0.141)
  Session 1: Lymphocytes, Day 7, n=2 | 0.05 (0.212)
  Session 1: Lymphocytes, Day 10, n=2 | -0.20 (0.424)
  Session 1: Lymphocytes, Day 26, n=2 | -0.10 (0.849)
  Session 2: Lymphocytes, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Lymphocytes, Day1-pre-dose, n=1 | -0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Lymphocytes, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Lymphocytes, Day 3, n=1 | -0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Lymphocytes, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Lymphocytes, Day 5, n=1 | -0.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Lymphocytes, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Lymphocytes, Day 7, n=1 | 0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Lymphocytes, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Lymphocytes, Day 10, n=1 | -0.40 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Lymphocytes, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Lymphocytes, Day 26, n=1 | -0.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Monocytes, Day 3, n=2 | 0.15 (0.212)
  Session 1: Monocytes, Day 5, n=2 | 0.10 (0.000)
  Session 1: Monocytes, Day 7, n=2 | 0.15 (0.212)
  Session 1: Monocytes, Day 10, n=2 | 0.15 (0.212)
  Session 1: Monocytes, Day 26, n=2 | 0.20 (0.141)
  Session 2: Monocytes, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Monocytes, Day1-pre-dose, n=1 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Monocytes, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Monocytes, Day 3, n=1 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Monocytes, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Monocytes, Day 5, n=1 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Monocytes, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Monocytes, Day 7, n=1 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Monocytes, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Monocytes, Day 10, n=1 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Monocytes, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Monocytes, Day 26, n=1 | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Neutrophils, Day 3, n=2 | 0.20 (0.707)
  Session 1: Neutrophils, Day 5, n=2 | 0.45 (1.202)
  Session 1: Neutrophils, Day 7, n=2 | 0.00 (0.000)
  Session 1: Neutrophils, Day 10, n=2 | -0.05 (0.212)
  Session 1: Neutrophils, Day 26, n=2 | 0.05 (0.354)
  Session 2: Neutrophils, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Neutrophils, Day1-pre-dose, n=1 | -0.70 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Neutrophils, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Neutrophils, Day 3, n=1 | -1.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Neutrophils, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Neutrophils, Day 5, n=1 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Neutrophils, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Neutrophils, Day 7, n=1 | -0.70 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Neutrophils, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Neutrophils, Day 10, n=1 | -1.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Neutrophils, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Neutrophils, Day 26, n=1 | 0.40 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Platelets, Day 3, n=2 | -7.5 (4.95)
  Session 1: Platelets, Day 5, n=2 | -29.5 (23.33)
  Session 1: Platelets, Day 7, n=2 | -21.0 (4.24)
  Session 1: Platelets, Day 10, n=2 | -13.0 (1.41)
  Session 1: Platelets, Day 26, n=2 | 12.0 (14.14)
  Session 2: Platelets, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Platelets, Day1-pre-dose, n=1 | -5.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Platelets, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Platelets, Day 3, n=1 | -32.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Platelets, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Platelets, Day 5, n=1 | -27.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Platelets, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Platelets, Day 7, n=1 | -31.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Platelets, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Platelets, Day 10, n=1 | -33.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Platelets, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Platelets, Day 26, n=1 | -9.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

69. Secondary Outcome: Part B: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: Blood samples were planned to be collected to analyze the hematology parameters.
Time Frame: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

70. Secondary Outcome: Part A: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: Hematocrit. Baseline was considered as the latest pre-dose assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Session 1: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26; Session 2: Day 1-Pre-dose, Days 3, 5, 7, 10 and 26
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Percentage of red blood cells in blood
  Session 1: Day 3, n=2 | -0.015 (0.0071)
  Session 1: Day 5, n=2 | -0.025 (0.0071)
  Session 1: Day 7, n=2 | -0.010 (0.0283)
  Session 1: Day 10, n=2 | -0.020 (0.0283)
  Session 1: Day 26, n=2 | -0.015 (0.0212)
  Session 2: Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Day1-pre-dose, n=1 | -0.040 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Day 3, n=1 | -0.040 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Day 5, n=1 | -0.040 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Day 7, n=1 | -0.050 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Day 10, n=1 | -0.040 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Day 26, n=1 | -0.050 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

71. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were planned to be collected to analyze the hematology parameter.
Time Frame: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

72. Secondary Outcome: Part A: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Hemoglobin. Baseline was considered as the latest pre-dose assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Session 1: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26; Session 2: Day 1- Pre-dose, Days 3, 5, 7, 10 and 26
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Grams per liter
  Session 1: Day 3, n=2 | -6.5 (2.12)
  Session 1: Day 5, n=2 | -10.5 (3.54)
  Session 1: Day 7, n=2 | -6.5 (3.54)
  Session 1: Day 10, n=2 | -8.0 (5.66)
  Session 1: Day 26, n=2 | -5.5 (2.12)
  Session 2: Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Day1-pre-dose, n=1 | -9.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Day 3, n=1 | -12.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Day 5, n=1 | -11.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Day 7, n=1 | -14.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Day 10, n=1 | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Day 26, n=1 | -17.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

73. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were planned to be collected to analyze the hematology parameter.
Time Frame: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

74. Secondary Outcome: Part A: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes Mean Corpuscular Hemoglobin. Baseline was considered as the latest pre-dose assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Session 1: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26; Session 2: Day 1- Pre-dose, Days 3, 5, 7, 10 and 26
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Picograms
  Session 1: Day 3, n=2 | 0.0 (0.00)
  Session 1: Day 5, n=2 | 0.0 (0.00)
  Session 1: Day 7, n=2 | 0.0 (0.00)
  Session 1: Day 10, n=2 | 0.5 (0.71)
  Session 1: Day 26, n=2 | 0.5 (0.71)
  Session 2: Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Day1-pre-dose, n=1 | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Day 3, n=1 | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Day 5, n=1 | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Day 7, n=1 | 1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Day 10, n=1 | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Day 26, n=1 | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

75. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were planned to be collected to analyze the hematology parameter.
Time Frame: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

76. Secondary Outcome: Part A: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes Mean Corpuscular Volume. Baseline was considered as the latest pre-dose assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Session 1: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26; Session 2: Day 1- Pre-dose, Days 3, 5, 7, 10 and 26
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Femtoliter
  Session 1: Day 3, n=2 | 0.75 (1.485)
  Session 1: Day 5, n=2 | 0.90 (0.707)
  Session 1: Day 7, n=2 | 1.85 (4.455)
  Session 1: Day 10, n=2 | 0.45 (1.061)
  Session 1: Day 26, n=2 | 0.60 (1.556)
  Session 2: Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Day1-pre-dose, n=1 | -2.60 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Day 3, n=1 | -2.50 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Day 5, n=1 | -3.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Day 7, n=1 | -0.90 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Day 10, n=1 | 1.50 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Day 26, n=1 | -0.90 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

77. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were planned to be collected to analyze the hematology parameter.
Time Frame: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

78. Secondary Outcome: Part A: Change From Baseline in Hematology Parameters: Erythrocytes, Reticulocytes
Description: Blood samples were collected to analyze the hematology parameters: Erythrocytes and Reticulocytes. Baseline was considered as the latest pre-dose assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Session 1: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26; Session 2: Day 1- Pre-dose, Days 3, 5, 7, 10 and 26
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
10^12 cells per liter
  Session 1: Erythrocytes, Day 3, n=2 | -0.175 (0.0212)
  Session 1: Erythrocytes, Day 5, n=2 | -0.295 (0.1485)
  Session 1: Erythrocytes, Day 7, n=2 | -0.180 (0.1556)
  Session 1: Erythrocytes, Day 10, n=2 | -0.230 (0.2687)
  Session 1: Erythrocytes, Day 26, n=2 | -0.200 (0.1273)
  Session 2: Erythrocytes, Day1-Pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Erythrocytes, Day1-Pre-dose, n=1 | -0.270 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Erythrocytes, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Erythrocytes, Day 3, n=1 | -0.340 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Erythrocytes, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Erythrocytes, Day 5, n=1 | -0.290 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Erythrocytes, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Erythrocytes, Day 7, n=1 | -0.480 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Erythrocytes, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Erythrocytes, Day 10, n=1 | -0.480 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Erythrocytes, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Erythrocytes, Day 26, n=1 | -0.470 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Reticulocytes, Day 3, n=2 | -0.0085 (0.00212)
  Session 1: Reticulocytes, Day 5, n=2 | -0.0085 (0.00636)
  Session 1: Reticulocytes, Day 7, n=2 | -0.0075 (0.00778)
  Session 1: Reticulocytes, Day 10, n=2 | -0.0065 (0.00919)
  Session 1: Reticulocytes, Day 26, n=2 | -0.0035 (0.01061)
  Session 2: Reticulocytes, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Reticulocytes, Day1-pre-dose, n=1 | -0.0100 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Reticulocytes, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Reticulocytes, Day 3, n=1 | -0.0180 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Reticulocytes, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Reticulocytes, Day 5, n=1 | -0.0140 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Reticulocytes, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Reticulocytes, Day 7, n=1 | -0.0100 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Reticulocytes, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Reticulocytes, Day 10, n=1 | -0.0170 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Reticulocytes, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Reticulocytes, Day 26, n=1 | -0.0030 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

79. Secondary Outcome: Part B: Change From Baseline in Hematology Parameters: Erythrocytes, Reticulocytes
Description: Blood samples were planned to be collected to analyze the hematology parameters.
Time Frame: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

80. Secondary Outcome: Part A: Change From Baseline in Chemistry Parameters: Glucose, Calcium, Potassium, Sodium, Urea
Description: Blood samples were collected to analyze the chemistry parameters: Glucose, Calcium, Potassium, Sodium and Urea. Baseline was considered as the latest pre-dose assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Session 1: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26; Session 2: Day 1- Pre-dose, Days 3, 5, 7, 10 and 26
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Millimoles per liter
  Session 1: Glucose, Day 3, n=2 | -2.40 (3.253)
  Session 1: Glucose, Day 5, n=2 | -2.45 (4.455)
  Session 1: Glucose, Day 7, n=2 | -3.25 (5.303)
  Session 1: Glucose, Day 10, n=2 | -3.60 (2.404)
  Session 1: Glucose, Day 26, n=2 | -2.60 (2.970)
  Session 2: Glucose, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Glucose, Day1-pre-dose, n=1 | 1.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Glucose, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Glucose, Day 3, n=1 | -1.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Glucose, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Glucose, Day 5, n=1 | -1.70 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Glucose, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Glucose, Day 7, n=1 | -2.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Glucose, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Glucose, Day 10, n=1 | -1.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Glucose, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Glucose, Day 26, n=1 | 0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Calcium, Day 3, n=2 | -0.050 (0.0141)
  Session 1: Calcium, Day 5, n=2 | -0.075 (0.0354)
  Session 1: Calcium, Day 7, n=1: number analyzed (Participants) | 1
  Session 1: Calcium, Day 7, n=1 | -0.090 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Calcium, Day 10, n=2 | -0.010 (0.1556)
  Session 1: Calcium, Day 26, n=2 | -0.030 (0.0424)
  Session 2: Calcium, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Calcium, Day1-pre-dose, n=1 | 0.020 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Calcium, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Calcium, Day 3, n=1 | -0.140 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Calcium, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Calcium, Day 5, n=1 | -0.030 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Calcium, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Calcium, Day 7, n=1 | -0.080 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Calcium, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Calcium, Day 10, n=1 | -0.040 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Calcium, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Calcium, Day 26, n=1 | 0.040 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Potassium, Day 3, n=2 | -0.10 (0.141)
  Session 1: Potassium, Day 5, n=2 | -0.10 (0.141)
  Session 1: Potassium, Day 7, n=1: number analyzed (Participants) | 1
  Session 1: Potassium, Day 7, n=1 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Potassium, Day 10, n=2 | -0.30 (0.141)
  Session 1: Potassium, Day 26, n=2 | -0.30 (0.000)
  Session 2: Potassium, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Potassium, Day1-pre-dose, n=1 | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Potassium, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Potassium, Day 3, n=1 | -0.50 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Potassium, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Potassium, Day 5, n=1 | 0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Potassium, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Potassium, Day 7, n=1 | -0.50 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Potassium, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Potassium, Day 10, n=1 | -0.40 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Potassium, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Potassium, Day 26, n=1 | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Sodium, Day 3, n=2 | 3.0 (1.41)
  Session 1: Sodium, Day 5, n=2 | -0.5 (0.71)
  Session 1: Sodium, Day 7, n=2 | 2.0 (1.41)
  Session 1: Sodium, Day 10, n=2 | 3.5 (0.71)
  Session 1: Sodium, Day 26, n=2 | 0.5 (3.54)
  Session 2: Sodium, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Sodium, Day1-pre-dose, n=1 | 1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Sodium, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Sodium, Day 3, n=1 | 4.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Sodium, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Sodium, Day 5, n=1 | 2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Sodium, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Sodium, Day 7, n=1 | 1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Sodium, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Sodium, Day 10, n=1 | 3.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Sodium, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Sodium, Day 26, n=1 | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Urea, Day 3, n=2 | 0.85 (1.202)
  Session 1: Urea, Day 5, n=2 | 1.00 (3.111)
  Session 1: Urea, Day 7, n=2 | -0.25 (1.344)
  Session 1: Urea, Day 10, n=2 | -0.20 (0.707)
  Session 1: Urea, Day 26, n=2 | 0.70 (1.273)
  Session 2: Urea, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Urea, Day1-pre-dose, n=1 | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Urea, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Urea, Day 3, n=1 | 1.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Urea, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Urea, Day 5, n=1 | 0.70 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Urea, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Urea, Day 7, n=1 | 0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Urea, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Urea, Day 10, n=1 | 0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Urea, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Urea, Day 26, n=1 | 0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

81. Secondary Outcome: Part B: Change From Baseline in Chemistry Parameters: Glucose, Calcium, Potassium, Sodium, Urea
Description: Blood samples were planned to be collected to analyze the chemistry parameters.
Time Frame: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

82. Secondary Outcome: Part A: Change From Baseline in Chemistry Parameters: Albumin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: Albumin and Protein. Baseline was considered as the latest pre-dose assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Session 1: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26; Session 2: Day 1- Pre-dose, Days 3, 5, 7, 10 and 26
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Grams per liter
  Session 1: Albumin, Day 3, n=2 | -2.0 (1.41)
  Session 1: Albumin, Day 5, n=2 | -2.0 (1.41)
  Session 1: Albumin, Day 7, n=2 | -1.0 (2.83)
  Session 1: Albumin, Day 10, n=2 | -2.0 (4.24)
  Session 1: Albumin, Day 26, n=2 | 0.5 (3.54)
  Session 2: Albumin, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Albumin, Day1-pre-dose, n=1 | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Albumin, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Albumin, Day 3, n=1 | -4.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Albumin, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Albumin, Day 5, n=1 | -4.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Albumin, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Albumin, Day 7, n=1 | -4.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Albumin, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Albumin, Day 10, n=1 | -6.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Albumin, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Albumin, Day 26, n=1 | -4.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Protein, Day 3, n=2 | -2.5 (0.71)
  Session 1: Protein, Day 5, n=2 | -6.0 (2.83)
  Session 1: Protein, Day 7, n=2 | -3.0 (1.41)
  Session 1: Protein, Day 10, n=1: number analyzed (Participants) | 1
  Session 1: Protein, Day 10, n=1 | -8.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Protein, Day 26, n=2 | 2.5 (9.19)
  Session 2: Protein, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Protein, Day1-pre-dose, n=1 | -3.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Protein, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Protein, Day 3, n=1 | -8.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Protein, Day 5, n=0: number analyzed (Participants) | 0
  Session 2: Protein, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Protein, Day 7, n=1 | -5.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Protein, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Protein, Day 10, n=1 | -7.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Protein, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Protein, Day 26, n=1 | -5.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

83. Secondary Outcome: Part B: Change From Baseline in Chemistry Parameters: Albumin, Protein
Description: Blood samples were planned to be collected to analyze the chemistry parameters.
Time Frame: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

84. Secondary Outcome: Part A: Change From Baseline in Chemistry Parameters: Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST)
Description: Blood samples were collected to analyze the chemistry parameters: ALP, ALT and AST. Baseline was considered as the latest pre-dose assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Session 1: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26; Session 2: Day 1- Pre-dose, Days 3, 5, 7, 10 and 26
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
International units per liter
  Session 1: ALP, Day 3, n=2 | -8.0984 (5.51433)
  Session 1: ALP, Day 5, n=2 | 0.2999 (17.39135)
  Session 1: ALP, Day 7, n=1: number analyzed (Participants) | 1
  Session 1: ALP, Day 7, n=1 | 7.7984 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: ALP, Day 10, n=2 | -2.0996 (2.96925)
  Session 1: ALP, Day 26, n=2 | -2.3995 (5.09015)
  Session 2: ALP, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: ALP, Day1-pre-dose, n=1 | 4.1992 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: ALP, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: ALP, Day 3, n=1 | 1.7996 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: ALP, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: ALP, Day 5, n=1 | 2.9994 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: ALP, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: ALP, Day 7, n=1 | -1.7996 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: ALP, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: ALP, Day 10, n=1 | -0.5999 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: ALP, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: ALP, Day 26, n=1 | 0.5999 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: ALT, Day 3, n=2 | -1.7647 (2.49569)
  Session 1: ALT, Day 5, n=2 | -3.5294 (4.99138)
  Session 1: ALT, Day 7, n=2 | -0.2941 (0.41595)
  Session 1: ALT, Day 10, n=2 | 1.1765 (1.66379)
  Session 1: ALT, Day 26, n=2 | -2.9412 (4.15948)
  Session 2: ALT, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: ALT, Day1-pre-dose, n=1 | 0.0000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: ALT, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: ALT, Day 3, n=1 | 0.0000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: ALT, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: ALT, Day 5, n=1 | 0.0000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: ALT, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: ALT, Day 7, n=1 | 0.0000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: ALT, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: ALT, Day 10, n=1 | 0.0000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: ALT, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: ALT, Day 26, n=1 | 0.0000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: AST, Day 3, n=2 | -5.3989 (4.24179)
  Session 1: AST, Day 5, n=2 | -7.1986 (7.63523)
  Session 1: AST, Day 7, n=2 | -3.2993 (1.27254)
  Session 1: AST, Day 10, n=2 | -2.9994 (0.84836)
  Session 1: AST, Day 26, n=2 | -3.2993 (5.51433)
  Session 2: AST, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: AST, Day1-pre-dose, n=1 | -0.5999 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: AST, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: AST, Day 3, n=1 | -5.3989 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: AST, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: AST, Day 5, n=1 | -4.7990 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: AST, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: AST, Day 7, n=1 | -4.1992 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: AST, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: AST, Day 10, n=1 | -5.3989 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: AST, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: AST, Day 26, n=1 | -4.1992 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

85. Secondary Outcome: Part B: Change From Baseline in Chemistry Parameters: ALP, ALT, AST
Description: Blood samples were planned to be collected to analyze the chemistry parameters.
Time Frame: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

86. Secondary Outcome: Part A: Change From Baseline in Chemistry Parameters: Direct Bilirubin, Bilirubin, Creatinine
Description: Blood samples were collected to analyze the chemistry parameters: Direct Bilirubin, Bilirubin, Creatinine. Baseline was considered as the latest pre-dose assessment prior to first administration of either study drug, i.e. GSK2315698 or anti-SAP mAb (labelled or unlabelled) (Day 1, Pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Session 1: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26; Session 2: Day 1- Pre-dose, Days 3, 5, 7, 10 and 26
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Micromoles per liter
  Session 1: Direct Bilirubin, Day 3, n=2 | -2.70 (2.121)
  Session 1: Direct Bilirubin, Day 5, n=2 | -4.35 (2.051)
  Session 1: Direct Bilirubin, Day 7, n=2 | -3.75 (3.323)
  Session 1: Direct Bilirubin, Day 10, n=2 | -2.80 (3.111)
  Session 1: Direct Bilirubin, Day 26, n=2 | -1.70 (0.707)
  Session 2: Direct Bilirubin, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Direct Bilirubin, Day1-pre-dose, n=1 | 0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Direct Bilirubin, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Direct Bilirubin, Day 3, n=1 | -0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Direct Bilirubin, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Direct Bilirubin, Day 5, n=1 | 0.60 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Direct Bilirubin, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Direct Bilirubin, Day 7, n=1 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Direct Bilirubin, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Direct Bilirubin, Day 10, n=1 | -0.50 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Direct Bilirubin, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Direct Bilirubin, Day 26, n=1 | -0.50 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Bilirubin, Day 3, n=2 | -9.30 (6.647)
  Session 1: Bilirubin, Day 5, n=2 | -12.30 (8.061)
  Session 1: Bilirubin, Day 7, n=2 | -11.85 (7.283)
  Session 1: Bilirubin, Day 10, n=2 | -9.55 (9.122)
  Session 1: Bilirubin, Day 26, n=2 | -5.10 (1.273)
  Session 2: Bilirubin, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Bilirubin, Day1-pre-dose, n=1 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Bilirubin, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Bilirubin, Day 3, n=1 | -2.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Bilirubin, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Bilirubin, Day 5, n=1 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Bilirubin, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Bilirubin, Day 7, n=1 | -1.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Bilirubin, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Bilirubin, Day 10, n=1 | -2.40 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Bilirubin, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Bilirubin, Day 26, n=1 | -2.70 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 1: Creatinine, Day 3, n=2 | 6.5 (6.36)
  Session 1: Creatinine, Day 5, n=2 | -4.5 (2.12)
  Session 1: Creatinine, Day 7, n=2 | 1.0 (0.00)
  Session 1: Creatinine, Day 10, n=2 | 1.0 (9.90)
  Session 1: Creatinine, Day 26, n=2 | 13.0 (1.41)
  Session 2: Creatinine, Day1-pre-dose, n=1: number analyzed (Participants) | 1
  Session 2: Creatinine, Day1-pre-dose, n=1 | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Creatinine, Day 3, n=1: number analyzed (Participants) | 1
  Session 2: Creatinine, Day 3, n=1 | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Creatinine, Day 5, n=1: number analyzed (Participants) | 1
  Session 2: Creatinine, Day 5, n=1 | -11.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Creatinine, Day 7, n=1: number analyzed (Participants) | 1
  Session 2: Creatinine, Day 7, n=1 | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Creatinine, Day 10, n=1: number analyzed (Participants) | 1
  Session 2: Creatinine, Day 10, n=1 | 1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2: Creatinine, Day 26, n=1: number analyzed (Participants) | 1
  Session 2: Creatinine, Day 26, n=1 | -2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

87. Secondary Outcome: Part B: Change From Baseline in Chemistry Parameters: Direct Bilirubin, Bilirubin, Creatinine
Description: Blood samples were planned to be collected to analyze the chemistry parameters.
Time Frame: Baseline (Day 1 Pre-dose), Days 3, 5, 7, 10 and 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

88. Secondary Outcome: Part A: Number of Participants With Abnormal Urinalysis Parameters: Glucose, Protein, Blood, Ketones
Description: Urine samples were collected to analyze urinalysis parameters including glucose, protein, blood and ketones.
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants | 2

89. Secondary Outcome: Part A: Number of Participants With Abnormal Urinalysis Parameters: Specific Gravity, Potential of Hydrogen
Description: Urine samples were collected to analyze urinalysis parameters including specific gravity and potential of hydrogen.
Time Frame: Up to Day 26 of the last session
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Anti-SAP
Number analyzed (Participants) | 2
Participants | 0

90. Secondary Outcome: Part B: Number of Participants With Abnormal Urinalysis Parameters: Glucose, Protein, Blood, Ketones
Description: Urine samples were planned to be collected to analyze the urinalysis parameters.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

91. Secondary Outcome: Part B: Number of Participants With Abnormal Urinalysis Parameters: Specific Gravity, Potential of Hydrogen
Description: Urine samples were planned to be collected to analyze the urinalysis parameters.
Time Frame: Up to Day 26
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Anti-SAP
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected up to Day 26 of the last session
Description: Safety population consisted of all participants who received at least one dose of GSK2315698, GSK2398852 or 89Zr-GSK2398852. AEs and SAEs were not collected in Part B as no participants were enrolled. Data is presented for Part A only as data was not collected in Part B due to the study was terminated during Part A, and Part B was not initiated.
Arm/Group | Part A: Anti-SAP
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Anti-SAP (N=2)
Headache (Nervous system disorders) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Injection site bruising (General disorders) | 1 (1)
Dactylitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT03417830/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT03417830/SAP_001.pdf